CLINICAL TRIAL: NCT03981510
Title: Comparison of Gastrointestinal Motility in Healthy Children and Children With Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3D-Transit Children AUH
Record Dates: First submitted 2019-06-07; First posted 2019-06-10 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-09

CONDITIONS: Constipation; Childhood Acute Lymphoblastic Leukemia; Neurofibromatosis 1; Chronic Constipation With Overflow
MeSH Terms: conditions — Constipation; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neurofibromatosis 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children being investigated with 3D-transit (Experimental): 4 groups of each 20 children will be investigated with respectively one or two capsules:
  * Healthy children (1)
  * Children with chronic constipation (2)
  * Children with neurofibromatosis type 1 (2)
  * Children with cancer receiving treatment with Vincristine (1)
  Interventions: Diagnostic Test: 3D-Transit

INTERVENTIONS:
Diagnostic Test: 3D-Transit — 3D transit investigation consists of a small electromagnetic pill and a detector located in a belt around the waist. The pill is swallowed by the participant and the belt is worn until the pill has left the gastrointestinal tract. The method is without any pain and discomfort for the child. The child will visit the hospital the first time to ingest the capsule alongside a standardized meal, and is then free to go home and proceed with daily activities (beside hard exersize) while wearing the belt with the detector. The next day, the child will again visit the hospital to check whether or not the capsule has left the tract - this is done with a computer and software. The children ingesting two capsules will do this with a certain delay.

SUMMARY:
To gain a better understanding of the underlying dysmotility in constipation in children, we will use a novel minimal invasive method called 3D Transit. We will examine four groups of children aged 7 to 17 years: healthy children, chronically constipated children (ROM IV criteria), children with neurofibromatosis type 1 and finally children receiving chemotherapy (vincristin) for acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria applicable to all participants:

• Children between 7-17 years of age where permission is granted for the participation by habitable parents with custody of the child. In case of joint custody, permission must be obtained from both parents.

Inclusion criteria applicable only to healthy participants:

• Gastrointestinal healthy children without chronic constipation

Inclusion criteria applicable only to constipated participants:

• Chronic constipation defined by Rom IV criteria, which is a diagnostic score for chronic constipation

Inclusion criteria applicable only to children in vincristine treatment:

• Children with cancer in treatment with vincristine

Inclusion criteria applicable only to patients with NF1:

• Diagnosis of NF1 with gastrointestinal symptoms

Exclusion Criteria:

* Children with parents who are unable to understand the given particpant's information
* Children with known dysregulated metabolic disease
* Previously major intra-abdominal surgery
* CNS surgery
* Other treatment-requiring gastrointestinal disorder
* Systemic steroid treatment within the last week
* Children with difficulty swallowing
* Children with known gastrointestinal obstruction or perforation
* Acute infections
* Diagnosed malabsorption including bile acid malabsorption
* Menarche in girls

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The investigation is without discomfort and adverse events. | 3 days
Children with chronic constipation has a longer transit time through the colon and fewer fast bowel movements than healthy children. | 3 days
Children in Vincristine treatment has a longer transit time through the colon and fewer fast bowel movements than healthy children. | 3 days
Children with NF1 and gastrointestinal symptoms has a longer transit time through the colon and fewer fast bowel movements than healthy children. | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Brinck CE, Mark EB, Ejerskov C, Johansen KB, Sutter N, Schlageter V, Drewes AM, Krogh K. Regional Gastrointestinal Motility in Healthy Children. J Pediatr Gastroenterol Nutr. 2021 Sep 1;73(3):306-313. doi: 10.1097/MPG.0000000000003198. PMID 34091540